CLINICAL TRIAL: NCT07343375
Title: Effect of High-intensity Interval Training on the Lung in Patients With COPD Referred for Lung Volume Reduction Surgery: The PREGENERATE Trial
Acronym: PREGENERATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Ronan Berg, MD, DMSc, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-25061713
Record Dates: First submitted 2025-12-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The HIIT intervention group includes three supervised sessions per week over the period while on waitinglist for lung volumen reduction surgery. These will take place at either CFAS or at home and will be supervised
  Interventions: Behavioral: High Intensity interval training (HIIT)
- Control group (No Intervention): Controls will be encouraged to maintain current exercise habits for the duration of the study.

INTERVENTIONS:
Behavioral: High Intensity interval training (HIIT) — The HIIT intervention consist of 4 intervals with each lasting 4 minutes (4x4min). If a participant reports discomfort related to the length of the intervals or start to feel unmotivated by performing the same exercise, we will use another HIIT protocol: 10x1min. The 4x4min HIIT consists of a warm-up period of 10 minutes with a target heart rate at 60-70% of HRmax, followed by 4 HIIT intervals with a target HR ≥85%. The intervals are separated by three minutes of active rest, in which the HR should drop to 60% of maximum. Following this, a cool down period of three minutes at warm up intensity is performed. The 10x1min HIIT consists of a 10-minute warm-up period.The warm-up is followed by 10 intervals, each lasting 1 min at 100% of maximal workload, separated by three minutes of active rest, in which the HR should drop to 60% of maximum. Following the intervals, a cool down period of three minutes at warm up intensity is performed.
  Arms: Exercise group

SUMMARY:
Patients with chronic obstructive lung disease (COPD) suffer from a progressive loss of lung function that leads to poor quality of life, and often invalidity and early death. Regular exercise can improve quality of life in these patients, but there is a lack in understanding the underlying mechanism of exercise-induced improvement in COPD and it is widely thought not to have any effect on the lung as such. In the present study, the investigators aim to investigate the impact of an extensive high-intensity interval training (HIIT)-based exercise scheme on the regenerative capacity of the lung in patients with COPD on waiting list for lung volume reduction surgery.

Design: Prospective randomized controlled clinical trial.

Intervention: 24 persons with COPD referred for lung volume reduction surgery will randomly be allocated (1:1) to prehabilitation with high intensity interval training (HIIT) or non-exercise control.

Outcomes: The primary outcome is differences in change in differential protein composition in distal lung tissue between HIIT and control groups post-intervention using spatial multimodal proteomics. Furthermore, lung tissue mass, protein composition (mass spectrometry and spatial omics e.g. MACSima), pulmonary blood volume, blood protein profile (biomarkers), diffusion capacity at rest and during exercise, oxygen consumption tests, body composition scan, distal airspace radii and physical functional tests will be measured before and after the intervention.

Perspective: This study may fundamentally change the view on the regenerative potential of the lungs in COPD.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) suffer from a progressive loss of lung function that leads to low physical performance, poor quality of life, and early death (2). Pulmonary rehabilitation, including exercise training, is considered the most effective non-pharmacological intervention for improving quality of life in patients with COPD (1). However, its use is halted by the lack of understanding of the mechanism of exercise-induced improvement in COPD, and is widely thought not to have any effect on lung function, at least as measured by dynamic spirometry and diffusion capacity measured at rest in the upright position (3,4). It is thus mainly considered a mean to alleviate symptoms, primarily by improving skeletal muscle function, but without the potential to reverse any structural changes within the pulmonary system which are seen in patients with COPD. The rationale for recommending exercise as a way to reduce symptom burden and increase quality of life, is based on the finding from the most recent Cochrane review (5). The authors stated that no additional studies comparing exercise with control were warranted, as exercise per se leads to improvements, regardless of the type of exercise.

The reasoning for not prescribing exercise more widely to patients with COPD is based on two assumptions: 1) new tissue cannot be formed in the adult lung, and 2) no consistent exercise training-induced changes in lung function have previously been documented.

However, de novo tissue formation has repeatedly been demonstrated in the adult lung, both in animals and humans, primarily in response to prolonged hypoxia and pneumonectomy (6,7). It has recently been reported that interval-based training counteracts the progressive loss of lung tissue in animal models of experimental COPD (8). The most likely stimulus is the mechanical strain, and if any measurable changes are to be induced by training, a high-intensity interval training (HIIT) scheme is preferable to be initiated in pulmonary rehabilitation (9).

An aspect of the progressive lung tissue loss in COPD that sets in from the very early stages of disease, seemingly before any ventilatory disturbance can be observed, is pulmonary vascular dysfunction and loss of pulmonary capillaries, driven by a seemingly disease-specific imbalance between angiogenetic and angiostatic processes in the pulmonary vasculature (10,11). Indeed, this is likely a mechanism that drives the concomitant loss of lung tissue, and also limits exercise capacity as the ability to expand the alveolar-capillary membrane though pulmonary capillary recruitment and distension becomes limited, thus critically attenuating oxygen uptake during exercise (10).

It is now well-established that the human lung conceals a diverse population of mechanosensitive progenitor and stem cells that appear to be dormant in COPD (12). Their reactivation by the stretch and strain as well as high vascular pressures associated with for example physical activity may likely explain why interval-based training has been found to counteract the progressive loss of lung tissue in animal models of experimental COPD (8,13,14). The investigators have developed in vitro protocols for assessing the regenerative capacity of the lung, and the next step will be to develop similar protocols for the human lung, both in the healthy state and from patients with COPD. In the present pilot study, the investigators will investigate the effects of an extensive high-intensity interval training (HIIT) on the regenerative capacity of the lung as determined by in vitro lung organoid culture and vascular tissue engineering 3D methods on patients with COPD on waiting list for lung volume reduction surgery.

Primary objective: To investigate whether prehabilitation with supervised HIIT while on waiting list for lung volume reduction surgery affects regenerative pathways in the lung. The investigators aim to determine if these effects can be detected non-invasively using blood biomarkers and spatial omics technologies to map region-specific molecular changes, cellular composition, and structural remodelling in lung tissue.

Secondary objectives: To determine whether an increase in blood volume is associated with an increased lung tissue mass (LTM), pulmonary blood volume (PBV), reduced symptom severity, and pulmonary diffusing capacity at rest and during exercise. To use explanted tissue to develop ex vivo models for disease and repair mechanisms (15,16).

Research hypotheses:

Primary: Prehabilitation while on waiting list for lung volume reduction surgery is superior to a non-exercise control group for increasing activating regenerative pathways in the lung with concomitant changes in LTM and PBV.

Secondary: Diffusing capacity during exercise and quality of life increases following prehabilitation with HIIT compared to a non-exercise control group. Finally, it is hypothesized that functional outcomes, V̇O2peak, body composition and cardiac output will be improved despite no/or limited changes in lung function in the HIIT group.

ELIGIBILITY:
Inclusion criteria

* Men and women
* Referred for lung volume reduction surgery at Rigshospitalet because of emphysematous COPD.

Exclusion criteria

* Symptoms of ischaemic heart disease
* Known heart failure
* Unable to complete or understand HIIT training
* Claudication
* Symptoms of acute disease within 2 weeks prior to the study
* Known malignant disease
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

  * Known chronic kidney or liver disease
  * Elevated creatinine, urea, alanine transaminase (ALAT), aspartate transaminase (ASAT), bilirubin, basic phosphatases at blood test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Differential protein composition | At surgery
  Differences in change in differential protein composition in distal lung tissue between HIIT and control group post-intervention using spatial multimodal proteomics.

SECONDARY OUTCOMES:
Differential protein composition | At surgery
  Differences in change in differential protein composition in distal lung tissue between HIIT and control group post-intervention using mass spectrometry.
Lung tissue protein composition | At surgery
  Differences in change in distal lung tissue protein composition pre- and post-HIIT intervention via mass spectrometry.
Serum protein profiles | At surgery
  Differences in change in serum protein profiles between HIIT and control groups after intervention using mass spectrometry.
Tissue niche and cellular composition | At surgery
  Tissue niche and cellular composition in the lung will be determined
Translational regions | At surgery
  Healthy, diseased and transitional (''border zones'') regions in the lung will be deliniated/identified by using spation omic analysis. This will be done both at a gene level, protein level and glycosaminoglycan level.
Inflammatory and remodelling factors (blood samples) | From time of inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in inflammatory and remodelling factor proteins in blood samples measured by mass spectrometry
Protein markers | At surgery
  Protein markers will be identified by mass spectrometry and the difference in the spatial localisation of these will be identified between the groups after the intervention. This will be done using Pentachrome and/or multiplexed inmunofluorescence stainings.
Lung cell population | At surgery
  Difference in change from baseline to follow-up between groups in lung cell populations by single cell-RNA sequencing.
Lung tissue mass | From inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in total LTM (g)
Pulmonary blood volume at rest | From inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in pulmonary blood volume (mL) at rest
DLNO at rest and during exercise | From inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in DL,NO (mmol/(min kPa)) as a function of V̇O2 measured at rest, 60% of current maximal workload (relative), and at follow-up including 60% of maximal workload at baseline (absolute)
DLNO during exercise | From inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in DL,NO (mmol/(min kPa)) during exercise at 60% of current maximal workload (relative)
DLNO during exercise | From inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in DL,NO (mmol/(min kPa)) during exercise at 60% of the maximal workload measured at baseline (absolute)
Pulmonary blood volume / total blood volume ratio | From inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in pulmonary blood volume / total blood volume ratio
Health related quality of life | From enrollment until 3 months post-surgery
  Difference in change from baseline to follow-up between groups in health-related quality of life - COPD Assessment Test (CAT) score, and St. George's Respiratory Questionnaire (SGRQ)
Extra cellular matrix structure | At surgery
  Extracellular matrix structure
Inflammatory and remodelling factors (lung tissue) | At surgery
  Difference in change from baseline to follow-up between groups in inflammatory and remodelling factor proteins in lung tissue measured by mass spectrometry

OTHER OUTCOMES:
Tissue morphology | At surgery
  Difference in change from baseline to follow-up between groups in tissue morphology
Mechanotransduction pathways | At surgery
  Detect increased activation of mechanotransduction pathways, marked by YAP/TAZ co-transcription factors, in lung tissue post-HIIT using spatial omics and advanced image analysis.
Mesenchymal stromal cells | At surgery
  Difference in mesenchymal stromal cells from baseline until follow-up between the two groups
Inflammatory patterns | At surgery
  Inflammatory patterns will be assessed understanding the difference in these inflammatory patterns from baseline until follow-up and the differences between the two groups
Distal airspace dimensions | From enrollment to surgery
  Difference in change from baseline to follow-up between groups in distal airspace dimensions (rAiDA and R0) as measured by AiDA
Neo-epitopes | At surgery
  Difference in change from baseline to follow-up between groups in neo-epitopes (degraded fragments of proteins) in lung tissue measured by mass spectrometry
Changes in X-ray and electron-based imaging techniques | At surgery
  Difference in change from baseline to follow-up between groups in elemental and structural changes by X-Ray and electron-based imaging techniques
Biophysical properties | At surgery
  Difference in change from baseline to follow-up between groups in biophysical properties (stiffness/elasticity) using tensile or atomic force microscopy (AFM
Lung function | At surgery
  Differences in above measurements linked to lung function
Cell activity | At surgery
  Differences in above measurements linked to cell activity
Lobal lung tissue mass | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in lobar LTM (g)
LTM/1.73 m2 BSA | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in LTM/1.73 m2 BSA (g/m2)
Total blood volume | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in total blood volume
DLNO during rest | From inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in DL,NO (mmol/(min kPa)) during upright rest
DLCOc during rest | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in DL,CO,5s (mmol/(min kPa)) during upright rest
Pulmonary capillary blood volume | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in pulmonary capillary blood volume (VC, mL) during upright rest
Membrane diffusing capacity | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in alveolar-capillary membrane diffusing capacity (DM, mmol/(min kPa)) during upright rest
Cardiac hemodynamics during exercise | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in cardiac output (L/min) during exercise at 60% of current maximal workload and 60% of baseline maximal workload, and during upright rest
VO2 during diffusing capacity measurements | From inclusion in the study until surgery (up to 8 months)
  DL,CO,NO-based V̇O2 during exercise at 60% of current maximal workload and 60% of baseline maximal workload, and during upright rest
Cardiac pulmonary exercise test outcomes | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in relative (mL/kg/min) V̇O2peak
Handgrip-strength | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in hand-grip strength (kg)
Sit-to-stand | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in numbers of completed 60 seconds sit-to-stand test (n)
Body composition | From inclusion in the study and until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in body composition: total mass (kg)
Lung function | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in lung function: FEV1 (L and %pred)
6-minutes walking distance | From enrollment until 3 months post surgery
  Difference in change in the distance (m) walked from baseline to follow-up between groups in a 6-minute walking test
Exercise-induced cytokine response | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in exercise-induced cytokine responses (interleukin-6 (pg/mL)
Mean bolus transit time - rest | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in mean bolus transit time (s) (supine rest)
Mean bolus transit time exercise | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in mean bolus transit time (s) (adenosine infusion)
Coronary flow reserve | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in global coronary flow reserve (mL/min)
Pulmonary blood volume reserve | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in pulmonary blood volume reserve (mL)
Ejection fraction | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in left ventricular ejection fraction (%)
Cardiac dynamics - rest | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in cardiac output (L/min) (supine rest)
Cardiac dynamics - exercise | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in cardiac output (L/min)
Total plasma volume | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in total plasma volume
Red blood cells | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in red blood cells
Coronary calcium score | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in coronary calcium score
Blood samples | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in blood samples: lipids (cholesterol (mmol/l)
Lung resistance | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in resistance (Rrs, R5-R20) measured by IOS
Lung reactance | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in reactance (Xrs, X5) measured by IOS
Cardiac function and structure | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in cardiac structure and function including
Progenitor cell changes | At surgery
  Difference in progenitor cells from baseline until follow-up between the two groups
Cardio pulmonary test outcomes | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in absolute (mL/min) V̇O2peak
Cardiac pulmonary exercise test outcomes | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between group in ventilatory threshold (%)
Cardiac pulmonary exercise test outcomes | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in ventilatory reserve (%)
Body composition | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in body composition: total fat mass (kg and %)
Body composition | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in body composition: lean body mass (kg)
Body composition | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in body composition: fat percentage (%)
Lung function | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in lung function: FVC (L and %pred)
Lung function | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in lung function: RV (L and %pred)
Lung function | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in lung function: , TLC (L and %pred)
Lung function | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in lung function: single-breath diffusion capacity to carbon monoxide (mmol/(min kPa) and %pred)
Exercise-induced cytokine response | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in tumour necrosis factor-α (pg/mL)
Exercise-induced cytokine response | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in C-reactive protein (μg/mL)
Exercise-induced cytokine response | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in interleukin-8 (pg/mL)
Exercise-induced cytokine response | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in interleukin-10 (pg/mL))
Cardiac dynamics - rest | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in heart rate (bpm) (supine rest)
Cardiac dynamics - rest | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in stroke volume (mL) (supine rest)
Cardiac dynamics - exercise | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in cardiac output (L/min) (adenosine infusion)
Cardiac dynamics - exercise | From inclusion in the study until surgery (up to 8 months)
  Difference in change from baseline to follow-up between groups in stroke volume (mL) (adenosine infusion)
Blood samples | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in blood samples: LDL (mmol/l)
Blood samples | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in blood samples: HDL (mmol/l))
Blood samples | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in blood samples: HbA1C (mmol/l)
Blood samples | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in blood samples: HsCRP (mg/L)
Blood samples | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in blood samples: pro-BNP (pmol/L)
Blood samples | From enrollment until 3 months post surgery
  Difference in change from baseline to follow-up between groups in blood samples: TSH (10-3 IU/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided